CLINICAL TRIAL: NCT04185155
Title: Preventing Intrusive Memories After Trauma Via a Simple Cognitive Intervention in the Hospital Emergency Department: "EKUT" (Enkel Kognitiv Uppgift Efter Trauma) - A Randomized Controlled Trial (RCT)
Brief Title: Simple Cognitive Task After Trauma EKUT RCT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Halted prematurely - Covid-19 pandemic prevented recruitment/testing in ED
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Emily Holmes, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-05380
Record Dates: First submitted 2019-11-28; First posted 2019-12-04 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple cognitive task (Experimental): A memory cue followed by playing the computer game "Tetris" on own smartphone. Options to engage in self-administered booster sessions after day 1.
  Interventions: Behavioral: Simple cognitive task
- Attention placebo (Placebo Comparator): Smartphone activity for same amount of time.
  Interventions: Behavioral: Attention placebo

INTERVENTIONS:
Behavioral: Simple cognitive task — A memory cue followed by playing the computer game "Tetris" on own smartphone. Options to engage in self-administered booster sessions after day 1.
  Arms: Simple cognitive task
Behavioral: Attention placebo — Smartphone activity for same amount of time.
  Arms: Attention placebo

SUMMARY:
This research study is designed to investigate the effects of a simple cognitive task (a memory cue following by playing the computer game "Tetris") on intrusive memories ("flashbacks") and other symptoms after a traumatic event. Patients presenting to a hospital emergency department soon after a traumatic event will be randomly allocated to either the simple cognitive task intervention or control. Participants will be followed up at one week and one month, and where possible 3 and 6 months. It is predicted that participants given the simple cognitive task intervention will develop fewer intrusive memories and less severe related clinical symptoms than those who are not. This will inform the future development of a simple technique to prevent distressing psychological symptoms after a traumatic event. Implementation and training aspects in a hospital context will also be explored. Patients use their smartphone for part of the intervention in the study.

DETAILED DESCRIPTION:
This is a Randomised Controlled Trial informed by prior feasibility and pilot work (ClinicalTrials.gov ID: NCT03509792). The primary outcome is the number of intrusive memories of the traumatic event (week 5). The intervention is delivered in emergency departments of Swedish hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Experienced or witnessed a traumatic event resulting in admission to the emergency department
* Met the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM5) criterion A for Posttraumatic Stress Disorder (PTSD) in that ("The person was exposed to actual or threatened death, serious injury, or sexual violence" by "Directly experiencing the traumatic event(s)" or "Witnessing, in person, the event(s) as it occurred to others")
* Can be seen in the emergency department ca. 6 hours after the traumatic event (day 1)
* Report memory of the accident
* Fluent in spoken and written Swedish
* Alert and orientated
* Have sufficient physical mobility to use their smartphone
* Willing and able to provide informed consent and complete study procedures
* Willing and able to be contacted following discharge to complete follow-up assessments
* Have access to an internet enabled smartphone

Exclusion Criteria:

* Loss of consciousness of > 5 minutes
* Current intoxication
* Report a history of severe mental illness
* Current substance abuse or neurological condition
* Currently suicidal
* Other medical reasons (on advice by medical staff)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Number of intrusive memories of traumatic event | Week 5
  Number of intrusive memories of traumatic event recorded by participants in a brief diary daily (morning, afternoon, evening and night) for 7 days.

SECONDARY OUTCOMES:
Number of intrusive memories of traumatic event | Week 1
  Number of intrusive memories of traumatic event recorded by participants in a brief diary daily (morning, afternoon, evening and night) for 7 days.
Impact of Event Scale - Revised (IES-R): Degree of subjective distress of post-trauma intrusion symptoms | One week and 1, 3, and 6 month follow-up
  Self-report measure that assesses subjective distress after a traumatic event (with reference to ED event). Here we include the intrusion subscale (8 items) and the avoidance subscale (8 items). Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Subscale scores are calculated for the Intrusion or Avoidance items summed (ranging from 0 to 32 each). Higher scores indicate worse outcome.
Hospital Anxiety and Depression Scale (HADS): Anxiety and depressive symptoms | One week and 1, 3, and 6 month follow-up
  The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. Higher scores indicate worse severity.
Posttraumatic Stress Disorder Checklist 5 (PCL-5) | One week and 1, 3, and 6 month follow-up
  Full scale is a 20-item self-report measure that assesses current symptoms of post-traumatic stress disorder. Items are rated on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). The PCL-5 yields a total symptom severity score which ranges from 0 to 80. Subscale symptom severity scores for DSM-5 symptom cluster B - intrusion symptoms (items 1-5), cluster C - avoidance (items 6-7), cluster D - negative alterations in cognitions and mood (items 8-14), and cluster E - alterations in arousal and reactivity (items 15-20). Higher scores indicate worse severity.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS) | One week and 1, 3, and 6 month follow-up
  A 12-item self-rated questionnaire measuring difficulties due to health conditions, including mental or emotional problems (with reference to ED study event). Scores range from 1 ("none") to 5 ("extremely/cannot do"). The maximum score of the WHODAS is 60, lower scores are better. 3 additional items measure on how many of the last 7 days (modified time scale) these difficulties occurred.

OTHER OUTCOMES:
Credibility/expectancy questionnaire | Day 1
  5 item questionnaire (11-point scale from 0 to 10) that rates to what degree the participants finds the intervention credible. High scores indicate greater credibility.
Subjective units of distress (SUDS) | Day 1
  A bespoke manipulation check item measuring self-rated distress during the intervention/control procedure (11-point scale from 0 to 10) at 3 times during the intervention process. Higher scores indicate higher level of distress.
Self-Rated initial intrusions | Day 1 and Day 2
  A question measuring the presence of intrusive memories with a yes/no response, and if yes then a free text response field to specify the number of intrusive memories and any comments, then 3 self rated items measuring the level of distress, vividness or concentration disruption associated with the intrusions (11 point scales from 0 to 10) given before intervention/control procedure in ED on day 1 and remotely on day 2.
Feedback Questionnaire about Participation | 1 month follow-up
  7 bespoke items including questions about study participation e.g. how acceptable was it to do the task at the emergency department? Rated on 11-point scale from 0 (not at all) to 10 (extremely), higher scores indicate higher acceptability; and questions about what has happened since the study with a yes/no response e.g. have you had any psychological or medical treatment since our last contact; and items with a free text response field e.g. do you have any other comments.
Self Rated Health (SRH) rating | Day 1, one week and 1, 3, and 6 month follow-up
  A single item measuring perceived health status on a seven-point scale (from very good to very bad). High scores indicate good outcomes.
Self Rated Sleep ratings | Day 1, one week and 1, 3, and 6 month follow-up
  Two self rated items: Item 1 measures the extent of being troubled by poor sleep (with reference to ED study event) on a 5 point scale (from not at all to very much), and item 2 measures the number of nights in the week with sleep problems on 5 point scale (from 0-1 to 5-7 nights). Each 5-point scale is reverse scored (0 - 4) then summed. Possible total scores range from 0 - 8, with higher values indicative of better sleep.
Characteristics of intrusive trauma memories | Week 1 and week 5, 3 and 6 month follow-up
  3 self rated items measuring the level of distress, vividness and concentration disruption associated with the intrusions (11 point scales from 0 to 10) rated within the diary at week 1 and 5 and in platform at 3 and 6 months. High scores indicate higher level of distress/vividness/concentration disruption.
Self Rated Functioning and social support ratings | One week, 1, 3, and 6 month follow up
  2 bespoke items including a question on impact on daily functioning associated with the intrusions and a question on perceived social support after the traumatic event. Both items are rated on an 11-point scale (from 0 "none"; 5 "some"; 10 "extreme/much"). High scores indicate higher level of functional impairment/perceived social support.
Intrusion questionnaire | One week and 1, 3, and 6 month follow-up
  6 self rated items measuring the frequency of unwanted memories of the trauma in the previous week on a 7-point scale (from never to many times a day) and the level of distress, nowness, reliving, disconnectedness and whether different triggers are associated with the unwanted memories of the trauma on a 11-point scale (from 0 to 100). High scores indicate more unwanted memories, higher levels of distress/nowness/reliving/disconnectedness and more different triggers.
Adverse events | One week and 1, 3, and 6 month follow-up
  A free text response field measuring the occurrence of any health problems since the last contact.
Training evaluation checklists | Through study completion, an average of 1 year
  To assess the researcher's training and adherence to study protocol. Uses competency items rated on a 7-point scale (from "absence" to "excellence", high scores indicate higher level of competency); factual questions as a yes/no response; and items with a free text response field for other feedback and comments.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Holmes, Prof, Principal Investigator — Karolinska Institutet/Uppsala University
Locations (1):
- Emergency Departments (e.g. FO Akut, Karolinska University Hospital Huddinge), Huddinge, Sweden

REFERENCES:
- [Result] Kanstrup M, Singh L, Goransson KE, Gamble B, Taylor RS, Iyadurai L, Moulds ML, Holmes EA. A simple cognitive task intervention to prevent intrusive memories after trauma in patients in the Emergency Department: A randomized controlled trial terminated due to COVID-19. BMC Res Notes. 2021 May 10;14(1):176. doi: 10.1186/s13104-021-05572-1. PMID 33971951